CLINICAL TRIAL: NCT06001580
Title: A Phase Ia Open-label, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Antitumor Activity of BR101 Injection, as a Single Agent in Subjects With Advanced Solid Tumors
Brief Title: A Study of BR101 Injection Alone in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioRay Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR101-I
Record Dates: First submitted 2023-08-04; First posted 2023-08-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BR101 (Experimental)
  Interventions: Drug: BR101

INTERVENTIONS:
Drug: BR101 — BR101 injection was administered once for 28 days observation period and then weekly until the subject experienced unacceptable toxicity, disease progression, poor compliance, pregnancy, informed withdrawal, death, study interruption, and withdrawal from the study

SUMMARY:
This study is a phase Ia study of single drug BR101 for Advanced solid tumor. The main purpose of this study is to Evaluate the safety and tolerability of BR101monotherapy (single dose and multiple doses) in Subjects with Advanced Solid Tumors and determine the MTD if possible, and determine the RP2D.

The secondary purpose of this study is to explore the Pharmacokinetics, Immunogenicity, Antitumor Activity of BR101 monotherapy (single dose and multiple doses) in Subjects with Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who voluntarily sign the informed consent form with an understanding of the nature, purpose and procedures of the trial, and can comply the protocol;
* 2. Males and females with an age of or above 18 years;
* 3. Patients with advanced or metastatic solid tumors diagnosed by pathological histology and / or cytology (cell wax only) who are unable for radical surgical resection, or who have failed to standard treatment or who have been intolerant to standard treatment (disease progression, or intolerant to chemotherapy, targeted therapy, etc.), or who lack effective treatment;
* 4. At least one measurable lesion according to RECIST V1.1;
* 5. ECOG score ≤ 1;
* 6. A recovery of previous treatment releated toxic reactions (except for the residual hair loss effect) to or under Grade 1 (according to CTCAE v 5.0) and a complete recovery of the immune-related adverse effects if the patients received anti-tumor treatment before;
* 7. Sufficient organ and bone marrow function;
* 8. The expected survival above 12 weeks;
* 9. Blood HCG test of females with a reproductive potential should be negative;
* 10. Fertile men and women must use a highly effective contraceptive methods, and continue the birth control for six months after the last dose.

Exclusion Criteria:

* 1. An current active autoimmune disease or history;
* 2. A history of primary immunodeficiency;
* 3. An current interstitial lung disease or history (except local interstitial lung disease induced by radiotherapy);
* 4. An active tuberculosis or history;
* 5. Any active infection that requires systemic treatment through intravenous infusion within 14 days before first dose;
* 6. Two or more primary tumors (excluding cured cervical in situ carcinoma, basal cell carcinoma or squamous cell skin cancer, and other tumors that have been treated and stable for more than 5 years);
* 7. Symptomatic or untreated metastasis in brain or other central nervous system. However, patients with CNS matastasis that has been completed removed and/or be stable or relieved after radiotherapy can be enrolled;
* 8. Uncontrollable pleural fluid, ascites, or pericardial effusion assesed by the investigator;
* 9. Patients with any of the following heart diseases: any grade of heart failure assesed by NYHA, severe cardiac arrhythmias requiring treatment, Unstable angina pectoris，myocardial infarction occurred within 3 months before the first dose, QTc≥480 ms, hypertension that cannot in good control, receiving PTCA or CABG within 6 months before the first dose;
* 10. Patients received anti-tumor therapy or participated in other clinical studies and used other test drugs 28 days before the first dose; Patients received the traditional Chinese medicine within 7 days before the first dose;
* 11. A history of psychopathy;
* 12. A history of major surgery or radiotherapy within 28 days before the first dose or expecting to operate a major surgery during the trial, a history of therapeutic radioactive agents within 56 days prior to the first dose;
* 13. A history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* 14. Patients who have a bleeding tendency or are receiving thrombolytic or anticoagulant therapy;
* 15. Patients who had been vaccinated within 28 days before the first dose or intend to be vaccinated during the trial;
* 16. Patients who had a history of blood donation within 3 months before the first dose, or plan to donate blood during the trial;
* 17. Patients who need to receive corticosteroids for more than 7 days (methylprednisolone > 10 mg/d or the equivalent dose) or other immunosuppressants within 14 days before the first dose, except for inhaled corticosteroids;
* 18. Patients with a positive presence in terms of antibody to human immunodeficiency virus should be excluded; patients with a positive treponema pallidum specific antibody test require a further testing of the treponema pallidum non-specific antibody, and if the result is also positive, the subject shoule be excluded; patients with a positive hepatitis C virus antibody test require a further testing of the hepatitis C virus RNA [HCV RNA], and if the result is also positive, the subject shoule be excluded; patients with a positive hepatitis B virus antibody test require a further testing of the hepatitis B virus DNA [HBV DNA], and if the result is also positive, the subject shoule be excluded;
* 19. Patients with diseases affecting intravenous injection and blood sample collection;
* 20. Pregnant or lactating women;
* 21. A plan to donate sperm from the signing of ICF to 6 months after the last dose;
* 22. A situation or a possibility that patients can't comply the protocal;
* 23. Other situations that are not suitable to attend this trial assesed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Safety, Tolerability,RP2D | up to 91 days after the last administration
  The incidence and severity of various adverse events of DLT, evaluated per NCI CTCAE 5.0 standard, abnormal physical examination, vital signs, laboratory examination, 12-guided ECG, etc.; maximum tolerated dose (MTD)(if possible).
  Recommended Phase II clinical trial dose

SECONDARY OUTCOMES:
Cmax | From screening to 31 days after the last administration
  Cmax
Tmax | From screening to 31 days after the last administration
  Tmax
AUC0-last | From screening to 31 days after the last administration
  AUC0-last
AUC0-tau | From screening to 31 days after the last administration
  AUC0-tau
Cmin | From screening to 31 days after the last administration
  Cmin
Immunogenicity assessment | From screening to 31 days after the last administration
  Anti-drug antibody (ADA) level produced by subjects
DCR | up to end of day 71
  DCR
DoR | up to end of day 71
  DoR
TTR | up to end of day 71
  TTR
CR | up to end of day 71
  CR
PFS | up to end of day 71
  PFS
Objective response rate(ORR) | up to end of day 71
  ORR
Pharmacodynamic assessment | UP to end of day 102
  After administration, to evaluate Total/free CD73 level in peripheral blood, CD73 enzymatic activity in peripheral blood, CD73 level and CD73 occupancy of peripheral blood T lymphocytes, CD73 level and CD73 occupancy of tumor tissue, CD73 enzymatic activity in tumor tissue, CD8+ tumor infiltrating lymphocyte level in tumor tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang, China